CLINICAL TRIAL: NCT04789629
Title: Effect of Low Level Laser Therapy on Hamstring Muscle Tightness and Calf Muscle Spasticity in Cerebral Palsy Children.
Acronym: cp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Laser Enhanced Sciences (Other)
Responsible Party: Principal Investigator, basma ragab, physiotherapist, National Institute of Laser Enhanced Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NILES; our team (Other: cairo universtity)
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: low level laser; spasticity; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Low-Level Light Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomize clinical trail
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level laser , physiotherapy (Active Comparator): Instrumentation Diode laser device will use for biostimulation of the muscle fiber . The device has a wavelength of 808 nm and a power output 0-250 mW. parameters of laser : Wavelength 808 nm Power output 100 mW Spot size 0.0314 cm2 Power density 3,18 W/cm2 Treatment time per point 40 s Energy density per point 4,77 J/cm2 Energy per point 4 J 12 sessions for one month with traditional physiotherapy ( stretching , strenghthing exercises , trunk control , balance training , standing exercises , gait training .)
  Interventions: Device: low level laser therapy
- physiotherapy (Active Comparator): traditional physiotherapy ( stretching , strenghthing exercises , trunk control , balance training , standing exercises , gait training ) for one hour
  Interventions: Device: low level laser therapy

INTERVENTIONS:
Device: low level laser therapy — 3 session per week laser with exercises
  Other Names: physiotherapy

SUMMARY:
Background :Spasticity is a motor disorder in children with cerebral palsy (CP) Cp is a non progress lesion in unmature brain lead to a group of chronic disorders that affect movement and posture development, may be accompanied by epilepsy, secondary musculoskeletal problems, deformaties and disturbances of sensation, perception, cognition, communication, and behavior Few studies demonstrate effectiveness of laser therapies in spasticity in cp.

Methodology : This study is randomize control trail aimes to evaluate the effect of low-level laser therapy (LLLT) on the spasticity of hamstring and calf muscle in children with CP over 12 session of intermittent laser exposures. Muscle tone , gross motor function, rang of motion (rom ) and poplital angle will evaluate before and after laser irradiation in 30 children with CP both geneder aged between two to six years old diaplegic clidren , exclusion children who take botox or done surgery . Muscles will irradiated with low-intensity diode laser pulses of 808-nm wavelength three times per week over one month follow up for one month.

DETAILED DESCRIPTION:
This is a randomized controlled study, in which the 30 children with diaplegic randomly divide into control and study groups by excel sheat on computer, each group include 15child. Each child will receive laser at a frequency of three sessions per week for 12 session, in addition to conventional physiotherapy program, while the control group have 15 child will receive conventional physiotherapy. Four variables will choose to detect the effect of laser therapy: (1) muscle tone, (2) range of motion (ROM) , (3) gross movement,(4) poplital angle assessment . These values will recorde in both groups before starting treatment and after the treatment period and after one month of stop treatment .

.

ELIGIBILITY:
Inclusion Criteria:

* spastic diaplegic children aged between 2 to 6years have spastic hamstring and calf muscle .

Exclusion Criteria:

* for post-operative children , children who take botox, children with contracture or fixed deformity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale | one month of treatment
  scale to assets muscle tone
Modified Ashworth scale | 2 months
  scale to assets muscle tone
rom by Goniometer | one month of treatment
  clinical assessment
rom by Goniometer | 2 months
  clinical assessment
poplital angle test | one month of treatment
  clinical test
poplital angle test | 2 months
  clinical test

SECONDARY OUTCOMES:
gross motor | one month of treatment
  GMFS88
gross motor | 2 months
  GMFS88

CONTACTS AND LOCATIONS:
Overall Officials: osama mr fekery, prof, Study Chair — NILES; asmaa ms osama, assist prof, Study Chair — physical therapy faculty; mostafa mr mohmed, bachaloria, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Out Clinic of Physical Therapy Faculty, Giza, El Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided